CLINICAL TRIAL: NCT07304557
Title: COMPARISON OF THE EFFECTS OF OROFACIAL AND TONGUE EXERCISES APPLIED AS AN ADDITION TO MYOFUNCTIONAL TREATMENT IN TEMPOROMANDIBULAR JOINT DISORDERS ON PAIN, JOINT AND TONGUE FUNCTIONS: A RANDOMIZED CONTROLLED TRIAL
Brief Title: Effects Exercises in Temporomandibular Joint Disorders on Pain, Joint and Tongue Functions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tayfun ISIK (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor-Investigator, Tayfun ISIK, Master of Science, Lecturer, Ankara Medipol University
Organization: Ankara Medipol University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0354; 0354 (Registry Identifier: IZMIR KATIP CELEBI UNIVERSITY HEALTH RESEARCH INSTITUONAL REVİEW BOARD)
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: TMD; TMD/Orofacial Pain
Keywords: Orofacial Pain; TMD; Tongue Strength; OMES
MeSH Terms: conditions — Facial Pain | interventions — Exercise; Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orofacial Group (Experimental): The group planned to orofacial exercises and manual therapy intervention applying.
  Interventions: Other: Exercise; Other: Manual therapy
- Control Group (Active Comparator): the group planned to manual therapy apply.
  Interventions: Other: Exercise; Other: Manual therapy

INTERVENTIONS:
Other: Exercise — The orofacial and tongue exercises include four-directional tongue mobilizations and resisted tongue movements in forward and upward directions within the oral cavity to improve tongue mobility. In addition, safe mouth opening exercises, as well as cheek and lip exercises, are also included in the exercise program.
  Other Names: Orofacial exercises; TMD exercises
  Arms: Orofacial Group
Other: Exercise — * Through in education program, participants will be informed about joint characteristics, eating and drinking habits, and behavioral training.
  * Diaphragmatic breathing will be taught to promote relaxation of the cervical muscles and to establish a proper breathing pattern.
  * Postural exercises will be instructed to improve neck and back mechanics.
  * Relaxation training may help reduce joint activity that increases during periods of stress.
  * When necessary, participants will also receive education on the appropriate use of hot and cold agents.
  Other Names: Home Exercise
Other: Manual therapy — Manual therapy will begin with cervical stretching, relaxation of the cervical paraspinal muscles, and release techniques for the sternocleidomastoid and scalene muscles.
  The intensity of these exercises will be adjusted according to the patient's and tissue's tolerance.
  Relaxation of the masticatory muscles will be achieved through massage applied externally to the jaw and the temporal region.
  Passive range-of-motion exercises will be performed to increase the mobility of the temporomandibular joint.

SUMMARY:
The goal of this clinical trial is to learn if orofacial exercises works to treat temporomandibular disorders in adults. It will also learn about the safety of orofacial exercises on temporomandibular disorders. The main questions it aims to answer are:

Does orofacial exercises improve function of temporomandibular disorders ? Does orofacial exercises decrease pain in temporomandibular disorders?

Researchers will compare orofacial exercises and manual therapy to manual therapy.

Participants will:

Take manual therapy and orofacial exercises or manual therapy two days in every week for 6 weeks Assessment once every 2 weeks for tests

DETAILED DESCRIPTION:
The study will be conducted with two groups. While the control group will receive myofunctional therapy, the intervention group will receive orofacial and tongue exercises in addition to myofunctional therapy. The inclusion of orofacial and tongue exercises in the intervention group constitutes the main hypothesis of the study. The myofunctional therapy consists of home exercises, normal cervical joint movements, and massage techniques targeting the masticatory muscles.

At baseline, participants' eligibility for inclusion will be assessed. Individuals who meet the inclusion criteria will be randomly assigned to one of the two groups using a sealed envelope randomization method. Evaluation of participants will begin with the collection of demographic data. After recording the demographic information, further assessments will be conducted through questionnaires and instrumental measurements.

The first assessment will focus on pain evaluation, using three different methods.

1. Numerical Pain Scale (NPS): This scale assesses pain intensity in three different conditions - during chewing, at rest, and during sleep. Participants will rate their pain on a scale from "0" (no pain) to "10" (worst imaginable pain).
2. Pain Catastrophizing Scale (PCS): This self-administered questionnaire evaluates the participant's thoughts and emotional responses related to pain.
3. Algometry: The pain thresholds of the superficial masticatory muscles (masseter and temporalis) will be determined. Three measurements will be taken from the most prominent point of each muscle with the algometer applied perpendicularly to the skin. The highest value among the three will be recorded as the pain threshold for that muscle.

Jaw function will be another measured parameter, assessed using two different methods-one questionnaire and one physical evaluation.

1. Jaw Functional Limitation Scale-20 (JFLS-20): This 20-item self-reported scale evaluates the functional limitations of the jaw and masticatory system. Higher scores indicate greater functional limitation.
2. Orofacial Myofunctional Evaluation with Scores (OMES): This protocol includes multiple subcomponents that assess facial and temporomandibular function, appearance, and range of motion.

Tongue strength and endurance will be measured using the same device. Participants will be seated upright in a chair during the assessment. Tongue strength will be evaluated in two parts - anterior and posterior.

* For anterior tongue strength, the device bulb will be positioned on the palate just behind the upper front teeth, and the participant will be asked to press it with the tongue.
* For posterior tongue strength, the bulb will be placed on the posterior palate, and the participant will press it with the middle part of the tongue.

Three measurements will be taken, and the highest value will be recorded as the maximal tongue strength.

Quality of life will be evaluated using a self-administered questionnaire - the Oral Health Impact Profile (OHIP) - which assesses the perceived impact of oral health on daily life.

After completing all baseline assessments, participants will receive the assigned intervention according to their group allocation. Regardless of group assignment, all participants will be given home exercises, which include patient education about the joint, eating and drinking habits, and behavioral training. Diaphragmatic breathing exercises will be taught to promote relaxation of cervical muscles and proper breathing patterns. Posture exercises will be included to improve neck and back mechanics. Relaxation training will be provided to help reduce joint overactivity during stress. Participants will also be instructed on the appropriate use of thermal agents (hot and cold packs) when needed.

Myofunctional therapy will begin with cervical stretching, relaxation of paraspinal cervical muscles, and release techniques for the sternocleidomastoid and scalene muscles. Exercise intensity will be adjusted according to the patient's tolerance and tissue response. Massage techniques targeting the masticatory muscles and the temporal region will be applied to promote relaxation. Passive range of motion exercises will be performed to increase temporomandibular joint mobility.

Orofacial and tongue exercises aim to improve tongue mobility and include four-direction tongue mobilizations, resisted forward and upward tongue movements, safe mouth opening exercises, as well as cheek and lip exercises.

The intervention program will consist of 12 sessions conducted twice a week for 6 weeks, with each session lasting approximately 45 minutes. Every two weeks, tongue strength and endurance, pain thresholds (via algometry), and pain levels (via NPS) will be reassessed.

Adherence to home exercises will be monitored at each session. Participants' compliance with both supervised and home exercise programs will be recorded using exercise logs.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 65 aged people
* Not having received physical therapy for the neck or jaw within the past three months.
* No history of surgical or oncological treatment related to the neck or jaw.
* Having a diagnosis of temporomandibular disorder according to the RDC/TMD criteria, specifically Group Ia, Group Ib, or Group IIa under Axis I.

Exclusion Criteria:

* Individuals who are pregnant or suspected to be pregnant.
* Individuals with rheumatologic diseases affecting the temporomandibular joint.
* Individuals with a diagnosed psychiatric disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
orofacial myofunctional evaluation with scores | From enrolment to the end of treatment at 6 weeks, in every two weeks
  The Orofacial Myofunctional Evaluation with Scores (OMES) protocol is designed to assess oral dysfunctions through multiple subdomains. These subdomains include appearance and posture, mobility, function, swallowing, mastication, functional occlusion, and mandibular movement. Higher scores indicate better functional status. The protocol has not yet been validated in Turkish. It was first used in a pediatric population and has also demonstrated validity in individuals with temporomandibular disorders.

SECONDARY OUTCOMES:
Pain threshold level of temporomandibular joint and temporal regions | From enrollment to the end of treatment at 6 weeks, once every two weeks.
  Pain thresholds will be measured using an algometer. In this study, the measurement sites are the masseter muscle (2.5 cm anterior and 1.5 cm inferior to the tragus) and the temporalis muscle (3 cm above the lateral edge of the eye). During the measurement, the algometer will be held perpendicular to the skin. Measurements will be conducted in a quiet room. Each site will be measured three times with 30-second intervals between measurements, and the average of the three measurements will be used for analysis. The validity of algometric measurements has been previously established.
Pain Level of Numerical Pain Scale | From enrollment to the end of treatment at 6 weeks, once in every two weeks
  The Numerical Pain Scale (NPS) is a self-reported or clinician-administered measurement tool that uses a numerical rating scale ranging from "no pain" to "worst possible pain". The scale is typically presented as a horizontal or vertical line and most commonly ranges from 0-10 or 0-100. It can be administered either in written or verbal form. Participants are asked to rate the intensity of their pain along this scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Medipol University, Ankara, ALTINDAG, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
A decision regarding the sharing of individual participant data (IPD) has not yet been made. The plan for data sharing will be evaluated as the study progresses and upon obtaining the necessary ethics approvals.